CLINICAL TRIAL: NCT03397966
Title: Metabolic Effects of Natriuretic Peptide Hormones
Acronym: MENP
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study drug no longer available
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: ENDA-025-17S; CX001678 (Other Grant/Funding Number: VA CSR&D)
Record Dates: First submitted 2017-12-20; First posted 2018-01-12 (Actual); Results first posted 2023-12-15 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Obesity; Cardiovascular Physiological Phenomena; Metabolism
Keywords: obesity; Cardiovascular Physiological Phenomena; metabolism; Energy Metabolism
MeSH Terms: conditions — Obesity | interventions — Natriuretic Peptide, Brain; Saline Solution

STUDY DESIGN:
Intervention Model Description: In this cross-over study, each subject will receive BNP infusion at one visit and placebo (control) at the other visit, in random order. The sequence of the treatments will be randomized. There will be a washout period (at least 14 days) between visits.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participant and study investigators will be blinded as to which infusion the participant is receiving at which visit. Also, the individuals analyzing the energy expenditure and fat gene expression will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- BNP, then placebo (Experimental): At Study Visit 1, subjects will receive an IV infusion of recombinant human b-type natriuretic peptide (BNP (1-32), nesiritide) for 240 minutes. After a washout period of at least 2 weeks, subjects then present for Study Visit 2, where they will receive an IV infusion of placebo (control, normal saline) for 240 minutes.
  Interventions: Drug: recombinant human BNP(1-32); Drug: placebo (control, normal saline)
- Placebo, then BNP (Experimental): At Study Visit 1, subjects will receive an IV infusion of placebo (control, normal saline) for 240 minutes. After a washout period of at least 2 weeks, subjects then present for Study Visit 2, where they will receive an IV infusion of recombinant human b-type natriuretic peptide (BNP (1-32), nesiritide) for 240 minutes.
  Interventions: Drug: recombinant human BNP(1-32); Drug: placebo (control, normal saline)

INTERVENTIONS:
Drug: recombinant human BNP(1-32) — Subjects will receive an IV infusion of recombinant human BNP(1-32) for 240 minutes at a rate of 10 ng/kg/minute for 240 minutes, preceded by an IV bolus of 100 ng/kg.
  Other Names: nesiritide, Natrecor
Drug: placebo (control, normal saline) — Subjects will receive an IV infusion of placebo (normal saline) at a rate of 10 ng/kg/minute for 240 minutes, preceded by an IV bolus of 100 ng/kg.

SUMMARY:
Accumulating evidence suggests that the natriuretic peptide (NP) hormonal system has important effects on metabolism. However, more information is needed to better understand the effects of NPs on metabolism in humans. Therefore, the investigators propose a study to determine the effects of b-type natriuretic peptide (BNP) on energy and fat metabolism in humans. The investigators' primary hypothesis is that the administration of BNP will increase energy expenditure in humans. The investigators' secondary hypothesis is that BNP administration will promote changes in gene expression in fat tissue suggestive of fat "beiging" in humans. Interventions that safely increase energy expenditure and promote fat "beiging" represent potential strategies for treating metabolic dysfunction due to obesity.

DETAILED DESCRIPTION:
Objective: The natriuretic peptide (NP) hormonal system is well-known for its important role in blood pressure regulation. However, accumulating evidence suggests that the NPs have significant effects on metabolism as well. For instance, administration of B-type natriuretic peptide (BNP) to wild-type mice leads to increased energy expenditure, changes in gene expression in fat tissue suggestive of fat "beiging" (which may be associated with cardiovascular and metabolic benefits), and reduced fat accumulation. Although recent studies in rodents suggest that NPs have important metabolic effects, there are few prospective data on the metabolic effects of NPs in humans.

Therefore, the investigators propose a physiologic, proof-of-concept study to determine the acute effects of b-type natriuretic peptide (BNP) on energy and fat metabolism in humans. The investigators' primary hypothesis is that the administration of BNP will increase energy expenditure in humans. The investigators' secondary hypothesis is that BNP administration will promote changes in gene expression in adipose tissue suggestive of a "beige" fat phenotype in humans.

Research Plan: The investigators propose the following research plan to address the investigators' specific aims:

Primary Aim: To investigate the acute effects of administration of BNP on energy expenditure in humans. The investigators propose a randomized, placebo-controlled, cross-over study in 50 adults (25 lean and 25 obese) without significant medical problems. Subjects will be randomized to intravenous infusion of recombinant human BNP(1-32) or normal saline (control), with assessment of energy expenditure and other physiologic measures. After a 7-day washout period, subjects will then undergo the other intervention.

Secondary Aim: To determine the acute effects of BNP on gene expression in white adipose tissue in humans. The investigators will assess markers suggestive of fat beiging in subcutaneous white adipose tissue biopsies after BNP infusion vs. control. This secondary aim will allow us to explore potential mechanisms underlying the hypothesized changes in energy expenditure.

Methods: In this cross-over study, each subject will receive BNP infusion at one visit and control at the other visit, in random order. The sequence of the treatments will be randomized. There will be a washout period (at least 14 days) between visits. Subjects will be stratified by BMI category (lean or obese). To address the Primary Aim, energy expenditure will be assessed via indirect calorimetry (metabolic cart). To address the Secondary Aim, subcutaneous fat biopsies will be performed, and tissue will be analyzed for gene expression of markers suggestive of fat beiging.

Clinical Relevance: This study will generate novel human data regarding the effects of the NPs on energy metabolism and adipose tissue. Interventions that safely increase energy expenditure and promote a beige fat phenotype represent potential strategies for treating obesity-associated metabolic dysfunction. The overarching scientific goals of this line of investigation are (1) to elucidate the role of the natriuretic peptide system in cardiometabolic health in humans, and (2) to investigate the potential for NP directed therapies in obesity-associated cardiometabolic dysfunction.

Update about Study Drug Supply Issues: The study started in 7/2018, and the last time participants were able to receive study drug was in May 2019, due to discontinuation of study drug by the drug manufacturer (nesiritide, Natrecor, Scios, LLC) after May 2019. Another potential source of drug supply was being sought out by the study team, and study recruitment was placed on hold during the search for new potential sources of study drug. A new viable source of study drug has not been identified, and funding is being closed. Thus, this study is being terminated. Results will be posted for the 5 participants who were able to complete the study procedures prior to the discontinuation of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18-40 years
* Body Mass Index (BMI): 18.5 BMI<25 kg/m2 (lean) or BMI > or = 30 kg/m2 (obese)

Exclusion Criteria:

* Significant cardiovascular disease (including heart failure and atrial fibrillation)
* Significant pulmonary, liver, or renal disease
* Diabetes Mellitus
* Significant Hypertension
* Hypotension
* Thyroid dysfunction
* Active malignancy
* Current or recent use of glucocorticoids
* Current use of antihypertensive medications, including diuretics
* Current use of medications affecting glucose metabolism, including metformin
* Current use of amphetamines or other medications known to affect energy homeostasis
* Currently pregnant or breastfeeding, or unwilling to avoid becoming pregnant or breastfeeding during study duration
* Significant claustrophobia that would prevent the use of the metabolic cart as part of the study protocol
* Currently abnormal serum or plasma sodium or potassium level
* Known hypersensitivity to recombinant human b-type natriuretic peptide, BNP(1-32) (nesiritide), or phenylephrine
* Hemoglobin A1c (HbA1c) >= 6.5%
* Liver Function Tests (LFTs) elevated >2x upper limit of normal
* Estimated Glomerular Filtration Rate (eGFR) <60 ml/min
* Currently abnormal thyroid stimulating hormone (TSH)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Talat A Ikizler, MD, Principal Investigator — Tennessee Valley Healthcare System Nashville Campus, Nashville, TN
Locations (2):
- United States (2):
  - Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Individual enrolled subjects will not receive any of their unique study data. IPD (in a de-identified, anonymized format) underlying publications from this research will be shared publicly.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Relevant IPA underlying a publication will be available within 6 months after publication date
Access Criteria: Data requests will be evaluated for appropriateness and relevance.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrolled subjects underwent a screening visit to determine eligibility for the study. The screening visit included a medical history, physical examination, and a blood draw for CMP, CBC, HbA1c, TSH, and free T4. A pregnancy test was completed on female subjects of child-bearing potential. Eligible subjects who still wished to participate in the study were then enrolled for the main study visits.
Groups:
- BNP Followed by Placebo (Control): At study visit 1, subjects will receive an IV infusion of recombinant human b-type natriuretic peptide (BNP (1-32)) for 240 minutes (at a rate of 10 ng/kg/minute, preceded by IV bolus of 100 ng/kg).
  After a washout of a minimum of 2 weeks, subjects will present for Study Visit 2, where they will receive an IV infusion of placebo control (normal saline) for 240 minutes.
- Placebo (Control) Followed by BNP: At study visit 1, subjects will receive an IV infusion of placebo (normal saline).
  After a washout of a minimum of 2 weeks, subjects will present for Study Visit 2, where they will receive an IV infusion of recombinant human b-type natriuretic peptide (BNP (1-32)) for 240 minutes (at a rate of 10 ng/kg/ minute, preceded by IV bolus of 100 ng/kg).
Period: Study Visit 1
Arm/Group | BNP Followed by Placebo (Control) | Placebo (Control) Followed by BNP
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0
Period: Washout Period (2+ Weeks)
Arm/Group | BNP Followed by Placebo (Control) | Placebo (Control) Followed by BNP
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0
Period: Study Visit 2
Arm/Group | BNP Followed by Placebo (Control) | Placebo (Control) Followed by BNP
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- BNP Followed by Placebo: At study visit 1, subjects will receive an IV infusion of recombinant human b-type natriuretic peptide (BNP (1-32)) for 240 minutes (at a rate of 10 ng/kg/minute, preceded by IV bolus of 100 ng/kg).
  After a washout of a minimum of 2 weeks, subjects will present for Study Visit 2, where they will receive an IV infusion of placebo control (normal saline) for 240 minutes.
- Placebo Followed by BNP: At study visit 1, subjects will receive an IV infusion of placebo (normal saline).
  After a washout of a minimum of 2 weeks, subjects will present for Study Visit 2, where they will receive an IV infusion of recombinant human b-type natriuretic peptide (BNP (1-32)) for 240 minutes (at a rate of 10 ng/kg/minute, preceded by IV bolus of 100 ng/kg).
- Total: Total of all reporting groups
Arm/Group | BNP Followed by Placebo | Placebo Followed by BNP | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 36 [28 to 38] | 34.5 [31 to 38] | 36 [31 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Resting Energy Expenditure (EE)
Description: At each visit (Study Visits 1 and 2), resting energy expenditure (EE) will be determined by indirect calorimetry, using a metabolic cart. Energy expenditure will be measured at baseline (just prior to the infusion) and during the 240-minute intravenous infusion at Study Visits 1 and 2. The primary endpoint will be change in resting energy expenditure, calculated as final resting energy expenditure (at end of 240-minute infusion) adjusted for baseline value.
Time Frame: At baseline and at end of 240-minute IV infusion (at each study visit). (At Study Visit 1 and 2, EE will be assessed at baseline and at end of 240-minute intravenous infusion. Visits will be separated by at least 14 days.)
Population: All participants who received both interventions and completed all study visits are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: kcal/day
Groups:
- BNP Infusion: Participants who received BNP infusion at either Study Visit 1 or Study Visit 2.
- Placebo (Control): Participants who received placebo (normal saline) infusion at either Study Visit 1 or Study Visit 2.
Arm/Group | BNP Infusion | Placebo (Control)
Number analyzed (Participants) | 5 | 5
kcal/day
  REE at baseline | 1867 [1649 to 1959] | 1800 [1769 to 2020]
  REE at end of infusion | 1970 [1687 to 1998] | 1883 [1782 to 1926]
Statistical Analysis 1: Comparison: BNP Infusion vs Placebo (Control); The primary endpoint is change in resting energy expenditure, calculated as final resting energy expenditure adjusted for baseline level, using linear regression. The null hypothesis is that there will be no significant effect of treatment on each endpoint. The investigators adhered to intention-to-treat principles. The test was performed with a significance level of 0.05; Test type: Superiority; p = 0.063, Mixed Models Analysis — The investigators tested the effect of treatment (BNP vs. control) on the primary endpoint using mixed effects modeling, adjusting for treatment sequence, to assess the effect of treatment on each endpoint

2. Secondary Outcome: Adipose Tissue Gene Expression of Uncoupling Protein 1 (UCP1)
Description: Subcutaneous adipose tissue biopsies will be obtained after the conclusion of the 240-minute IV infusion at Study Visits 1 and 2. These tissues will be analyzed for adipose tissue gene expression. The adipose tissue gene expression after the BNP infusion will be compared to expression after the placebo infusion. Units are relative UCP1 gene expression (quantified using quantitative real-time reverse-transcription polymerase chain reaction (qRT-PCR)), normalized to a housekeeping gene).
Time Frame: A subcutaneous biopsy will be collected after the end of 240-minute IV infusion, at both Study Visits 1 and 2 (Visits will be separated by at least 14 days.)
Population: All participants (N= 4) who had paired adipose tissue samples available (who had adipose tissue sample collected after both the BNP infusion and after the placebo infusion). There was 1 subject who did not have adipose tissue collected at one of the study visits, and thus is not included in the statistical analysis.
Measure: Mean (Standard Error); unit: fold change
Arm/Group | BNP Infusion | Placebo (Control)
Number analyzed (Participants) | 4 | 4
fold change | 9.66 (3.42) | 3.30 (1.18)
Statistical Analysis 1: Comparison: BNP Infusion vs Placebo (Control); The null hypothesis is that there will be no significant effect of BNP on adipose gene expression of UCP1 compared with placebo. The alternative hypothesis is that UCP1 expression would be significantly higher after BNP treatment compared with placebo; Test type: Superiority; p = 0.07, t-test, 2 sided — Paired t-test

ADVERSE EVENTS:
Time Frame: Approximately 1 year
Groups:
- BNP Followed by Normal Saline (Control): Subjects will initially receive an IV infusion of recombinant human b-type natriuretic peptide (BNP (1-32)) for 240 minutes. After a wash out of a minimum of 2 weeks subject will receive an IV infusion of normal saline for 240 minutes.
  recombinant human BNP (1-32): Subjects will receive an IV infusion of recombinant human BNP1-32 (6 mcg BNP/ml saline) for 240 minutes.
  normal saline (placebo): Subjects will receive an IV infusion of normal saline for 240 minutes. The volume of saline delivered will be equivalent to the volume of saline that the subject receives during the BNP infusion visit.
- Normal Saline (Control) Followed by BNP: Subjects will initially receive an IV infusion of normal saline for 240 minutes. After a wash out of a minimum of 2 weeks subject will receive an IV infusion of recombinant human b-type natriuretic peptide (BNP (1-32)) for 240 minutes. The volume of saline delivered will be equivalent to the volume of saline that the subject receives during the BNP infusion visit.
  normal saline (placebo): Subjects will receive an IV infusion of normal saline for 240 minutes. The volume of saline delivered will be equivalent to the volume of saline that the subject receives during the BNP infusion visit.
  recombinant human BNP (1-32): Subjects will receive an IV infusion of recombinant human BNP1-32 (6 mcg BNP/ml saline) for 240 minutes.
Arm/Group | BNP Followed by Normal Saline (Control) | Normal Saline (Control) Followed by BNP
All-Cause Mortality (participants affected / at risk) | 3/5 | 2/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 3/5 | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BNP Followed by Normal Saline (Control) (N=5) | Normal Saline (Control) Followed by BNP (N=5)
Local skin reaction (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) — Bruising at biopsy site.
Vasovagal response (Cardiac disorders) | 0 (0) | 1 (2) — Vasovagal response during biopsy.
Finger Fracture prior to intervention (unrelated to study) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Finger fracture occurred at home after screening visit and prior to receiving any intervention. Unrelated to study.
Headache (Vascular disorders) | 1 (1) | 0 (0) — Headache during study infusion.
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Nausea during study infusion.

LIMITATIONS AND CAVEATS:
Sample size is limited due to discontinuation of study drug (recombinant human BNP(1-32), nesiritide, Natrecor) by the drug manufacturer (Scios, LLC) after 5/2019. Results are posted for the 5 participants who were able to complete the study procedures prior to the discontinuation of study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-21): https://cdn.clinicaltrials.gov/large-docs/66/NCT03397966/Prot_SAP_000.pdf
  • Informed Consent Form (2018-12-27): https://cdn.clinicaltrials.gov/large-docs/66/NCT03397966/ICF_001.pdf